CLINICAL TRIAL: NCT05720468
Title: Exercise for Cognitive Excellence in Parkinson's Disease
Acronym: EXCEL-PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23NS123506 (NIH); K23NS123506 (NIH)
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise (Experimental): Participants randomized to the exercise group will receive 26 weeks of home-based, combined endurance and resistance training program under guidance and virtual supervision from exercise trainers. Exercise will be performed 5 days per week, with 3 days of endurance training using treadmill and 2 days of resistance training.
  Interventions: Other: Exercise
- Waitlist Control Group (Placebo Comparator): The control group will continue usual level of physical activity the participants were doing prior to enrollment in the study. At the end of the 26 week study period, participants will be offered the chance to participate in the same home-based, combined endurance and resistance training program.
  Interventions: Other: No Exercise

INTERVENTIONS:
Other: Exercise — Combined endurance and resistance exercise training
  Arms: Exercise
Other: No Exercise — Continue usual level of physical activity; option to participate in exercise training program after 26-week intervention period
  Arms: Waitlist Control Group

SUMMARY:
This study will evaluate the safety and feasibility of a home-based, virtually-supervised, combined high intensity endurance and resistance training program in people with Parkinson's disease. It will also evaluate the effects of exercise on cognition and underlying exercise-related biological markers (biomarkers).

DETAILED DESCRIPTION:
Cognitive impairment begins early in Parkinson's disease (PD) and progresses to dementia in a majority of patients, impairing quality of life and contributing to growing health-related costs. Physical exercise has potent anti-aging effects and improves many outcomes in PD including cognition. Identifying biomarkers that respond to exercise, and how they associate with cognition and underlying disease pathology, may elucidate key mechanisms for countering cognitive decline. This is a randomized-controlled trial that evaluates safety and feasibility of a home-based exercise intervention in people with PD and measure its effects on cognition and circulating biomarkers of aging and stress. Thirty-two participants with PD will be randomized to receive a home-based, trainer-supervised endurance and resistance training program (exercise group) or no exercise (wait list control group) for 26 weeks. Cognitive assessments and patient reported outcomes will be obtained at baseline and at end of 26 weeks. Biomarkers in periphery (blood, saliva) and brain [cerebrospinal fluid (CSF)] will also be measured before and after the 26-week exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic Parkinson's disease (PD) based on MDS criteria, with bradykinesia plus one of the other cardinal signs of PD (resting tremor, rigidity), without any other known or suspected cause of parkinsonism.
2. Modified Hoehn and Yahr stage less than 4
3. Age 40-80 years at time of screening
4. If being treated with PD symptomatic medications (i.e.g., rasagiline, carbidopa/levodopa, dopamine agonists, amantadine, anti-cholinergics), stable doses for greater than or equal to 2 months prior to baseline. If not being treated with PD symptomatic medication at time of screening, deemed unlikely to require symptomatic medication for next 6 months.

Exclusion Criteria:

1. A diagnosis of atypical parkinsonism, drug-induced parkinsonism, essential tremor, primary dystonia or other diagnoses that explain symptoms other than PD.
2. A diagnosis of a significant neurological disease other than PD that would interfere with ability to perform study procedures or assessments.
3. Significant cognitive impairment defined as Montreal Cognitive Assessment (MoCA)<23 or any impairment that would, in the opinion of the investigator, interfere with ability to follow exercise directions.
4. Beck Depression Inventory II (BDI) score > 16, indicating depression that precludes ability to exercise.
5. Use of neuroleptics/dopamine receptor blockers for more than 30 days in the year prior to baseline visit, or any use within 30 days of baseline visit.
6. Recent use of psychotropic medications (e.g., recent use of psychotropic medications (i.e., anxiolytics, hypnotics, benzodiazepines, antidepressants) where dosage has not been stable for more than 30 days prior to screening.
7. Presence of known cardiovascular, metabolic, or renal disease or individuals with major signs or symptoms suggestive of cardiovascular, metabolic, or renal disease without medical clearance to participate in the exercise program.
8. Presence of any of the following laboratory abnormalities on screening labs:

   1. Abnormal liver function (AST or ALT more than 2 times the upper limit of normal)
   2. Abnormal renal function (creatinine clearance calculated by the Cockcroft-Gault equation <50mL/min or estimated glomerular filtration rate using the MDRD4 equation or the CKD-EPI equation <45mL/min/1.73m2)
   3. Complete Blood Count out of range on screening labs and physician's judgment that abnormal value is clinically significant.
9. Uncontrolled hypertension (resting blood pressure >150/90 mmHg).
10. Orthostatic hypotension and standing systolic BP below 100. Orthostatic hypotension is a reduction of systolic blood pressure of at least 20 mm Hg or diastolic blood pressure of at least 10 mm Hg within 3 minutes of standing.
11. Already participating in 120 minutes or more of moderate intensity exercise per week.
12. Serious illness (requiring systemic treatment and/or hospitalization) within the last 4 weeks.
13. History of any other medical problem or injury that may interfere with ability to exercise.
14. Condition that precludes the safe performance of routine lumbar puncture, including:

    1. INR > 1.4 or other coagulopathy
    2. Platelet cell count of < 50,000/μL
    3. Infection at the desired lumbar puncture site
    4. Taking anti-coagulant medication within 90 days of baseline (Note: low dose aspirin is permitted)
    5. Suspected non-communicating hydrocephalus or intracranial mass
    6. Prohibitive lumbar spinal disease
15. Enrollment in another investigational study that includes an intervention; participation in non-interventional studies may be permitted
16. Receipt of any non-PD investigational product or device or participation in a non-PD drug research study within a period of 30 days (or 5 half-lives of the drug, whichever is longer) before baseline.
17. History of frequent falls (i.e. falling multiple times per week) or considered high fall risk based on investigator assessment
18. Lack of access to computer/tablet and WiFi or any other technical challenges that in the opinion of the investigator would prevent participation in the virtually supervised exercise training program.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Average percent heart rate maximum (HR max) | From weeks 5-26, every exercise session
  The overall average percent HR max will be compared to the target percent HR max (80-85 percent).
Average repetition maximum | From weeks 5-26, every exercise session
  The overall average repetition maximum for resistance exercise will be compared to the target repetition maximum (10-repetition maximum)
Average number of days per week exercised | From weeks 5-26, every week
  The average number of days per week exercised will be compared to target adherence (5 days/week of exercise)

SECONDARY OUTCOMES:
Change in cognitive function | Baseline and 26 weeks
  Change from baseline in Montreal Cognitive Assessment (MoCA). MoCA scores range between 0 and 30, with higher scores representing a better outcome.
Change in motor symptoms of Parkinson's disease | 26 weeks
  Change from baseline in the Movement Disorders Society-Unified Parkinson Disease Rating Scale motor score (Part III). The minimum score on the MDS-UPDRS Part III is 0 and the maximum is 132 with higher scores representing worse motor symptoms.
Change in biomarker of aging | Baseline and 26 weeks
  Change from baseline in blood levels of klotho
Change in biomarker of aging | Baseline and 26 weeks
  Change from baseline in CSF levels of klotho
Change in biomarker of stress | Baseline and 26 weeks
  Change from baseline in saliva levels of cortisol
Change in biomarker of stress | Baseline and 26 weeks
  Change from baseline in CSF levels of cortisol
Change in biomarker of inflammation | Baseline and 26 weeks
  Change from baseline in blood levels of CRP
Change in biomarker of inflammation | Baseline and 26 weeks
  Change from baseline in CSF levels of CRP
Change in neurotrophic biomarker | Baseline and 26 weeks
  Change from baseline in blood levels of BDNF
Change in neurotrophic biomarker | Baseline and 26 weeks
  Change from baseline in CSF levels of BDNF

OTHER OUTCOMES:
Change in isokinetic strength | Baseline and 26 weeks
  Change from baseline in maximal knee extension measured in peak torque
Change in isokinetic strength | Baseline and 26 weeks
  Change from baseline in handgrip strength measured in kilograms using dynamometer
Change in fitness | Baseline and 26 weeks
  Change from baseline in maximal oxygen consumption measured with peak oxygen volume
Change in walking capacity | Baseline and 26 weeks
  Change from baseline in distance in 6-minute walk
Change in quality of life | Baseline and 26 weeks
  Change from baseline in quality of life measured with the Parkinson Disease Questionnaire-39 (PDQ-39). The PDQ-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality over the last month covering 8 dimensions scored on a 5 point ordinal system (0=never, 4=always). Dimension score = sum of scores of each item in the dimension divided by the maximum possible score of all the items in the dimension, multiplied by 100. Each dimension total score range from 0 (never have difficulty) to 100 (always have difficulty). Lower scores reflect better QoL. Overall score can be summarized in the Parkinson's Disease Summary Index (PDSI) or PDQ-39 Summary Index (PDQ-39 SI).PDSI or PDQ-39 SI = sum of dimension total scores divided by 8.
Change in mood | Baseline and 26 weeks
  Change from baseline in mood measuring using the Beck Depression Inventory (BDI-II). The BDI-II is a 21-item self-report inventory designed to measure the severity of depression symptomatology. Each item is evaluated on a severity scale ranging from 0-3, with a total score ranging from 0-63. A score of 0-13 is considered none or minimal range depression; 14-19 mild is considered mild depression; 20-28 is considered moderate depression and 29-63 is considered severe depression.
Change in cognitive function | Baseline and 26 weeks
  Change from baseline in the National Institute of Health Toolbox Cognitive Battery, a comprehensive, performance-based test comprised of motor, emotion, sensation, and cognition assessments. For the purpose of this study, the investigators will be using the cognitive battery to assess processes involved in learning and comprehension (i.e. thinking, remembering, problem-solving, judging). The battery consists of tasks involving the use of executive function, memory, attention, and language.
Change in cognitive function | Baseline and 26 weeks
  Change from baseline in alternate phonemic/semantic fluency test. This test measures executive cognitive function. Participants are required to alternate letter-cued words with category-cued words. Higher scores represent a better outcome.
Change in cognitive function | Baseline and 26 weeks
  Change from baseline in Trail Making Test. This test is commonly used for the evaluation of attentional processes and cognitive flexibility. The Trail Making Test contains two components. The first part only demands simpler attentional processes - seeking numbers spread throughout a page, while the second involves a flexibility component requiring the participant to switch between numbers and letters during the test run. Higher scores represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nijee Luthra, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No